CLINICAL TRIAL: NCT05078515
Title: Multicenter Validation of the PREDICT Score for Prediction of Local Recurrence After Total Mesorectal Excision of Rectal Cancer
Brief Title: Multicenter Validation of the PREDICT Score
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Associate professor of surgery, Mansoura University
Other Study IDs: Mansoura2020110
Record Dates: First submitted 2021-10-02; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with recurrence after TME: Patients who developed local recurrence after TME of rectal cancer
  Interventions: Diagnostic Test: PREDICT score
- Patients without recurrence after TME: Patients who did not develop local recurrence after TME of rectal cancer
  Interventions: Diagnostic Test: PREDICT score

INTERVENTIONS:
Diagnostic Test: PREDICT score — Predictive score for local recurrence after TME for rectal cancer that includes 8 parameters

SUMMARY:
Even after adequate TME with grade III mesorectal grading, local recurrence remains a possible event. Several studies investigated different parameters and assessed their predictive power in regards to local recurrence after TME. These parameters included a variety of patient-related, tumor-related, and treatment-related factors. A recent meta-analysis reviewed the current literature for the predictors of local recurrence after TME for rectal cancer and developed a prognostic scoring system, the PREDICT score.

The present study aimed to validate the PREDICT scoring system by applying it to a prospective cohort of patients with rectal cancer who underwent curative TME in three

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex with non-metastatic low or middle rectal cancer who underwent elective TME with curative intent

Exclusion Criteria:

* Patients with recurrent or metastatic rectal cancer at the time of presentation
* Patients with synchronous colon cancer
* Patients with missing data on the outcome of TME.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-III rectal cancer who underwent surgery with curative intent
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of PREDICT score | 36 months after surgery
  The ability of the score to predict actual cases of recurrence after TME
Specificity of PREDICT score | 36 months after surgery
  The ability of the score to predict patients who did not experience recurrence after TME

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., FACS, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No